CLINICAL TRIAL: NCT06163664
Title: Role of ChatGPT in Vestibular Schwannoma Management
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was witbdrawn due to funding and resource limitations.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Janet Choi, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UP-23-00541
Record Dates: First submitted 2023-10-24; First posted 2023-12-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Vestibular Schwannoma
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention with 1 week use of ChatGPT
  Interventions: Behavioral: Use of chatGPT for 1 week
- Delayed control (Active Comparator): No ChatGPT use for 1 week and intervention after 1 week
  Interventions: Behavioral: Use of chatGPT for 1 week

INTERVENTIONS:
Behavioral: Use of chatGPT for 1 week — Use of chatGPT for 1 week

SUMMARY:
Previous studies have demonstrated that patients frequently undergo significant decision conflict regarding major medical decisions in otolaryngology. There lack validated tools available for decision support for patients. While limited evidence has demonstrated that clinical decision support tools can alleviate decision conflict for patients with diagnosis in otolaryngology, conversational language models were not employed in these studies and may provide additional benefit in this context. This study seeks to evaluate the efficacy of using ChatGPT, a conversational language model with basic clinical knowledge, in alleviating decision conflict for patients with new diagnosis in otolaryngology. For this pilot study, vestibular schwannoma, a benign tumor that develops on the vestibular nerve with known clinical equipoise, has been chosen for the initial study diagnosis. Efficacy will be evaluated by comparison of responses to the Decisional Conflict Scale (DCS) and Satisfaction with Decision (SWD) scores between a group given training in ChatGPT and a control group (no ChatGPT training).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosed with vestibular schwannoma
* Have access to internet-enabled device that is compatible with ChatGPT

Exclusion Criteria:

* < 18 years old
* patient without diagnosis of vestibular schwannoma
* patient does not have access to internet-enabled device
* patient who declines study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in scores of Decisional Conflict Scale after ChatGPT use | baseline, 1 week follow up, 2 week follow up
  The Decisional Conflict Scale (DCS) measures 5 dimensions of decision making (feeling: uncertain, uninformed, unclear about values, unsupported; ineffective decision making). 15-item validated questionnaire. Score range 5-75 (higher score corresponding to higher levels of conflict in decision making)
Changes in scores of Satisfaction with Decision after ChatGPT use | baseline, 1 week follow up, 2 week follow up
  The Satisfaction with Decision (SWD) scale measures satisfaction with health care decisions. 6-item validated questionnaire. Score range 5-30 (higher score corresponding to higher levels of satisfaction with decision)
Changes in scores for Knowledge on vestibular schwannoma management after ChatGPT use | baseline, 1 week follow up, 2 week follow up
  4-item questionnaire (Likert scale) assessing participants' confidence in understanding the diagnosis and treatment options for vestibular schwannoma. Score range 5-20 (higher score corresponding to higher levels of confidence in understanding diagnosis and management of vestibular schwannoma)

IPD SHARING:
Plan to Share IPD: Undecided